CLINICAL TRIAL: NCT01411306
Title: Screening for Swallowing Problems in Patients Following Prolonged Intubation: Validation of the Toronto Bedside Swallowing Screening Test (TOR-BSST©)
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 110957
Record Dates: First submitted 2011-08-04; First posted 2011-08-08 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Med/Surg ICU Inpatients, Intubated ≥ 48 hours
  Interventions: Other: Toronto Bedside Swallowing Screening Test (TOR-BSST©); Procedure: Videofluoroscopic Swallow Study

INTERVENTIONS:
Other: Toronto Bedside Swallowing Screening Test (TOR-BSST©) — All enrolled patients will be screened for dysphagia by two blinded screeners using the TOR-BSST©.
Procedure: Videofluoroscopic Swallow Study — All enrolled patients will undergo a videofluoroscopic assessment of swallowing within 24 hours of being screened with the TOR-BSST©.

SUMMARY:
Despite medical advances, half of the patients admitted to hospital for recovery from acute illness, injury or surgery have swallowing difficulties and those requiring tubes for breathing support are at even greater risk. Difficulties with swallowing decrease patients' quality of life, prolong their hospital stay, as well as lead to medical complications such as pneumonia, malnutrition and death. Presently, there is no screening test for swallowing difficulties in patients who have required respiratory support. Screening will allow for early detection of swallowing problems which is important to prevent serious complications, such as pneumonia. This research will determine the accuracy of a new screening test, the Toronto Bedside Swallowing Screening Test (TOR-BSST©) previously tested with stroke patients, to predict the presence of swallowing difficulties in patients who have required breathing support for longer than 48 hours. The investigators will enroll 100 patients from the intensive care medical surgical units at the University Health Network. The findings from this research will help identify those patients with swallowing problems earlier than it is currently possible. Once identified, at risk patients will be referred to a speech language pathologist swallowing expert for more comprehensive testing; thereby, decreasing their risk of experiencing serious complications, such as pneumonia, secondary to swallowing problems.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18+ years
* Inpatient at University Health Network, in any of the medical-surgical intensive care units, regardless of disease type, comorbidities or previous medical history
* Received endotracheal intubation lasting 48 hours or longer

Exclusion Criteria:

* History of one or more of the following: neurological disorder, surgery to the head or neck, previous oropharyngeal dysphagia, tracheotomy in situ or dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Med/Surg ICU inpatients who have received endotracheal intubation lasting 48 hours or longer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-05; Primary Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Validity of the TOR-BSST© | 24 hours
  The validity of the TOR-BSST© will be measured using sensitivity, specificity, likelihood ratios, positive predictive value (PPV), and negative predictive value (NPV). Results of the videofluoroscopic assessment of swallowing will be used as the gold standard comparison.
Inter-rater reliability of the TOR-BSST© | 24 hours
  Inter-rater reliability will be calculated using the intraclass correlation coefficient (ICC).

SECONDARY OUTCOMES:
Estimation of the incidence of dysphagia in adult acute patients following prolonged intubation | 24 hours
Description of the impairment characteristics of dysphagia in adult acute patients following prolonged intubation | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary Martino, PhD, Principal Investigator — University of Toronto / University Health Network
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] Barker J, Martino R, Reichardt B, Hickey EJ, Ralph-Edwards A. Incidence and impact of dysphagia in patients receiving prolonged endotracheal intubation after cardiac surgery. Can J Surg. 2009 Apr;52(2):119-24. PMID 19399206
- [Background] Martino R, Silver F, Teasell R, Bayley M, Nicholson G, Streiner DL, Diamant NE. The Toronto Bedside Swallowing Screening Test (TOR-BSST): development and validation of a dysphagia screening tool for patients with stroke. Stroke. 2009 Feb;40(2):555-61. doi: 10.1161/STROKEAHA.107.510370. Epub 2008 Dec 12. PMID 19074483
- [Background] Skoretz SA, Flowers HL, Martino R. The incidence of dysphagia following endotracheal intubation: a systematic review. Chest. 2010 Mar;137(3):665-73. doi: 10.1378/chest.09-1823. PMID 20202948
- [Background] Heffner JE. Swallowing complications after endotracheal extubation: moving from "whether" to "how". Chest. 2010 Mar;137(3):509-10. doi: 10.1378/chest.09-2477. No abstract available. PMID 20202944
- See also: Related Info — http://swallowinglab.uhnres.utoronto.ca/